CLINICAL TRIAL: NCT05434364
Title: Comparison the Effects of Facilitated Tucking, Swaddling and Prone Position Applied During Endotracheal Aspiration on Pain, Comfort and Physiological Parameters in Preterm Infants
Brief Title: Comparison Three Methods on Endotracheal Aspiration in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Kilis 7 Aralik University (Other)
Responsible Party: Principal Investigator, SERAP ÖZDEMİR, Doctor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IstanbulS
Record Dates: First submitted 2022-06-21; First posted 2022-06-28 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Preterm; Pain, Acute; Physiological Stress; Nursing Care; Comfort
MeSH Terms: conditions — Premature Birth; Acute Pain | interventions — Facilitated Tucking; Prone Position

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Facilitated Tucking (Experimental): giving facilitated tucking before, during and after the procedure
  Interventions: Other: Facilitated Tucking
- Swaddling (Experimental): giving swaddling before, during and after the procedure
  Interventions: Other: Swaddling
- Prone position (Experimental): giving prone position before, during and after the procedure
  Interventions: Other: Prone Position
- control (No Intervention): Rutin care in the neonatal intensive care unit

INTERVENTIONS:
Other: Facilitated Tucking — giving facilitated tucking before (1st and 3th minutes), during and after (1st and 3th minutes) the procedure
  Arms: Facilitated Tucking
Other: Swaddling — swaddling before (1st and 3th minutes), during and after (1st and 3th minutes) the procedure
  Arms: Swaddling
Other: Prone Position — giving prone position before (1st and 3th minutes), during and after (1st and 3th minutes) the procedure
  Arms: Prone position

SUMMARY:
Stress and pain control are vital for newborns, especially preterm babies. While painful procedures cause physiological changes in the short term, they negatively affect brain development in the long term. Non-pharmacological interventions with proven efficacy include: fetal position, sucrose, breastfeeding, breast milk, maternal presence, non-nutritive sucking, swaddling (wrapping) and skin-to-skin contact, as well as developmentally supportive positioning. Evaluating the effectiveness of nursing practices to be performed on babies, scientifically proving the most beneficial application that will both alleviate pain and increase their comfort in painful procedures such as aspiration and being more beneficial to babies are among the most basic benefits. Thanks to these applications, it is predicted that your baby will experience less pain and provide more comfort. Therefore, this study aim to comparison the effects of facilitated tucking, swaddling and prone position applied during endotracheal aspiration on pain, comfort and physiological parameters in preterm infants.

DETAILED DESCRIPTION:
The universe of the research; between July-September 2022, patients who are intubated on a mechanical ventilator at 32-36 weeks of gestation (middle preterm group) in Gaziantep Cengiz Gökçek Obstetrics and Pediatrics Hospital Neonatal Intensive Care Unit will consist of. In order to determine the sample size of the study, power analysis was performed using the G*Power (V3.1.9.7) program. According to Cohen's effect size coefficients; Assuming that the effect size (f = 0.4) of the evaluations to be made between four independent groups will be large/large, Taplak and Bayat (2021) found the effect size as 0.932 as a result of the Power analysis based on the PIPP-R results. In this study, it was determined that there should be at least 15 people in all groups (Fetal position, Swaddling, Prone position and control group) according to the new calculation made with 0.932 effect size, 5% alpha (two-sided) and 99% power. Considering that there may be losses during the study, each group will form a sample of 100 infants, 25 infants each. Random assignment of babies to groups will be carried out by the researcher through a computer program (https://www.randomizer.org)/. After determining the groups of premature babies randomly, one group will be given fetal position, one group swaddling position and one group prone position before, during and after endotracheal aspiration. Pain scores (PIPP-R), comfort scores (Comfort Scale) and physiological parameters (Heart peak beat, oxygen saturation value measured by pulse oximetry) 3 minutes before, during and after these nursing practices in the 1st and 3rd minutes after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Having 28-35 weeks of gestation,
* Follow-up as intubated in SIMV mode on mechanical ventilator,
* Follow-up on a ventilator between 1-10 days,
* Having a body weight of ≥1000 g,
* Those who have not taken any opioid or sedative medication until 4 hours before the procedure will be included.

Exclusion Criteria:

* Presence of congenital anomaly,
* Chest tube inserted
* Intracranial bleeding,
* Presence of condition/anomaly that will prevent prone tilting,
* Those with a history of epileptic seizures will be excluded.

Ages: 28 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-02-03 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Pain scores | 6 minutes
  Premature infant pain profile-revised (PIPP-R) (min=0 max=21, the higher the score, the more severe the pain)
Comfort score | 6 minutes
  Newborn Comfort Behavior Scale (min=6 max=30, High scores signify that the infant is not comfortable)
physiological parameter (Heart rate) | 6 minutes
physiological parameter (oxygen saturation) | 6 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Taplak AS, Bayat M. Psychometric Testing of the Turkish Version of the Premature Infant Pain Profile Revised-PIPP-R. J Pediatr Nurs. 2019 Sep-Oct;48:e49-e55. doi: 10.1016/j.pedn.2019.06.007. Epub 2019 Jun 19. PMID 31229348
- [Background] Hartley KA, Miller CS, Gephart SM. Facilitated tucking to reduce pain in neonates: evidence for best practice. Adv Neonatal Care. 2015 Jun;15(3):201-8. doi: 10.1097/ANC.0000000000000193. PMID 26002861
- [Background] Lopez O, Subramanian P, Rahmat N, Theam LC, Chinna K, Rosli R. The effect of facilitated tucking on procedural pain control among premature babies. J Clin Nurs. 2015 Jan;24(1-2):183-91. doi: 10.1111/jocn.12657. Epub 2014 Jul 24. PMID 25060423